CLINICAL TRIAL: NCT06612242
Title: Early vs. Late Tracheostomy in Patients With Guillain -Barre Syndrome: Comparison of Clinical Outcomes- a Retrospective Study
Brief Title: Early vs. Late Tracheostomy in Patients With Guillain -Barre Syndrome
Status: Recruiting | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Other Study IDs: 0206-24-MMC
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Guillain Barre Syndrome; Mechanical Ventilation
MeSH Terms: conditions — Guillain-Barre Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early tracheostomy: Patients with Guillain Barre who underwent early tracheostomy
  Interventions: Procedure: early tracheostomy (less than 7 days from intubation)
- Late tracheostomy: Patients with Guillain Barre who underwent late tracheostomy
  Interventions: Procedure: Late tracheostomy (more than 7 days from intubation)

INTERVENTIONS:
Procedure: early tracheostomy (less than 7 days from intubation) — Early tracheostomy (less than 7 days from ventilation) in mechanically ventilated patients with Guiilain-Barre syndrome
  Groups: Early tracheostomy
Procedure: Late tracheostomy (more than 7 days from intubation) — Late tracheostomy (more than 7 days from ventilation) in mechanically ventilated patients with Guiilain-Barre syndrome
  Groups: Late tracheostomy

SUMMARY:
Tracheostomy is one of the most common procedures in the intensive care unit in patients who need prolonged invasive mechanical ventilation. There is controversy in the literature regarding the ideal timing for performing tracheostomy in critically ill patients. Early tracheostomy may be associated with a decrease in ventilation days and hospitalization. We would like to investigate whether in ventilated patients with Guillain Barre syndrome, early tracheostomy will be associated with decreased ventilation days, decreased mortality and shorter hospital and ICU length of stay.

ELIGIBILITY:
Inclusion Criteria: All patients aged 18--99 who were admitted to the general intensive care unit from January 2012 to September 2024 with a diagnosis of Guillain-Barre syndrome who required mechanical ventilation and underwent tracheostomy during ICU stay.

-

Exclusion Criteria: Missing recoreded data

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 18--99 who were admitted to the general intensive care unit from January 2012 to September 2024 with a diagnosis of Guillain-Barre syndrome who required mechanical ventilation and underwent tracheostomy during ICU stay
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
ventilation days | 1 year from intubation
  number of ventilation days

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: Undecided